CLINICAL TRIAL: NCT04818853
Title: COVID-19 Associated Pulmonary Aspergillosis (CAPA) and Other Invasive Fungal Infections (IFI)
Acronym: CAPA IFI
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Peter Pappas, Principle Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300006311; 2023948 (Other Grant/Funding Number: Astellas); 2023158 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Covid19; Aspergillosis; Fungal Infection
Keywords: COVID19; Aspergillosis; Fungal; CAPA
MeSH Terms: conditions — COVID-19; Aspergillosis; Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Discarded clinical samples from routine testing will be collected and tested for diagnostic purposes on a weekly basis. These will include serum, deep suction specimens, and BAL when available. These samples will be tested for Aspergillus GM, Aspergillus PCR, and Pneumocystis PCR. Specimens will be stored at the CDC biorepository for future diagnostic use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID Patients with Aspergillosis and Other fungal Infections: All patients have been diagnosed with COVID-19. The purpose of this study is to look at this group of patients in the potential to develop Aspergillosis and other fungal infections.
  Interventions: Other: Observation to monitor patients for these infections

INTERVENTIONS:
Other: Observation to monitor patients for these infections — We will be receiving discarded specimens weekly. From these we are going to identify these various potential infections.

SUMMARY:
The purpose of this study is to identify the number of individuals with severe CoVID who require ventilator support and who develop serious fungal infections. The study is an observational study, meaning that we are not providing any intervention that does not involve usual standard of care. Our chief goal is to find evidence of fungal infection by using traditional, approved methods of diagnosis, but by applying these methods in the same way and frequency among all study participants. We will be looking especially for evidence of a fungal infection known as Aspergillus, which can causes a serious lung infection called invasive aspergillosis (IA).

DETAILED DESCRIPTION:
COVID-19 is a disease caused by infection with the novel coronavirus SARS-COV2 which emerged in late 2019 in Wuhan, China (1). This illness is associated with viral prodromal symptoms, then subsequently fever, cough, and shortness of breath (1). In a subset of patients, lower respiratory tract infection associated with respiratory failure develops. Among these patients, progression to severe respiratory failure and ARDS requiring ventilator support has occurred in an alarming number of patients at rates that are many-fold higher than what is typically associated with seasonal influenza A or B (2). One of the most feared complications of post-influenza respiratory failure is the development of invasive pulmonary aspergillosis which may occur in as many as 15-20% of those requiring ventilator support (based on European data) (3-6). Among those developing IA following influenza A or B, mortality of 50% or greater is reported (3-6).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older at the time of enrollment
* SARS-COV2 positivity by PCR with respiratory failure requiring mechanical ventilation for at least 72 hours
* Prior therapy with antifungals, including prophylaxis, is NOT an exclusion.

Exclusion Criteria:

* Life expectancy of less than 72 hours as determined by the site investigator.
* Expected to be weaned from mechanical ventilation in next 24 hours
* Care received in any setting other than an intensive care unit (ICU) at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Intensive Care Unit Patients with SARS-CoV2 requiring greater than 72 hours of mechanical ventilation.
  Participating sites include: University of Alabama at Birmingham, University of Pittsburgh, Washington University in St. Louis, University of California at Davis, University of Texas at Houston, University of Maryland, and University of Texas Health Sciences Center at San Antonio, Cornell University and Columbia/Presbyterian Medical Center
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Participants requiring mechanical ventilation | 72 hours or greater
  Number of patients placed on a ventilator
Participants with all cause mortality | In 30 days
  Participants with all cause mortality in SARS-CoV-2
Participants with all cause mortality | In 60 days
  Participants with all cause mortality in SARS-CoV-2

SECONDARY OUTCOMES:
Participants at risk for developing CAPA or IFIs | 180 days
  Risk factors associated with patients who are at risk for CAPA or IFIs

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pappas, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To Be Determined